CLINICAL TRIAL: NCT05808595
Title: A Randomized, Double-blind, Placebo Controlled, Parallel Clinical Trial to Investigate the Efficacy of AlphaWave® L-Theanine on Adults Who Experience Moderate Stress on a Regular Basis
Brief Title: The Safety and Efficacy of AlphaWave® L-Theanine on Adults Who Experience Moderate Stress on a Regular Basis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ethical Naturals, Inc. (Other)
Collaborators: KGK Science Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 22ENCLR01
Record Dates: First submitted 2023-03-17; First posted 2023-04-11 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2023-09

CONDITIONS: Stress
Keywords: Safety and efficacy; Stress

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AlphaWave® L-Theanine (Experimental): Participants will be instructed to take one capsule twice daily, once in the morning and once in the evening with water with or without food, starting on Day 1. If a dose is missed participants are instructed to take the missed dose immediately once noticed unless it is noticed within two hours of taking their next dose in which case, participants are instructed to document the missed dose and continue with their regular dosing schedule. Participants will be advised not to exceed 3 capsules daily.
  Interventions: Dietary Supplement: AlphaWave® L-Theanine
- Placebo (Placebo Comparator): Participants will be instructed to take one capsule twice daily, once in the morning and once in the evening with water with or without food, starting on Day 1. If a dose is missed participants are instructed to take the missed dose immediately once noticed unless it is noticed within two hours of taking their next dose in which case, participants are instructed to document the missed dose and continue with their regular dosing schedule. Participants will be advised not to exceed 3 capsules daily.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: AlphaWave® L-Theanine — One capsule of AlphaWave® L-Theanine will be taken twice daily for 28 days.
  Arms: AlphaWave® L-Theanine
Other: Placebo — One capsule of Placebo will be taken twice daily for 28 days.
  Arms: Placebo

SUMMARY:
The objective of this study is to evaluate the efficacy of AlphaWave® L-Theanine on stress among adults who experience moderate stress on a regular basis. The difference in change in stress as assessed by salivary cortisol from baseline at Days 14 and 28 will be compared between AlphaWave® L-Theanine and Placebo groups. Additionally, the safety and tolerability of AlphaWave® L-Theanine, as compared to placebo, will be measured by the occurrence of an/or changes in pre-emergent and post-emergent adverse events (AEs).

ELIGIBILITY:
Inclusion Criteria:

1. Males and females between 18 and 65 years of age, inclusive
2. Female participant is not of child-bearing potential, defined as females who have undergone a sterilization procedure (e.g. hysterectomy, bilateral oophorectomy, bilateral tubal ligation, total endometrial ablation) or have been post-menopausal for at least 1 year prior to screening Or,

   Females of child-bearing potential must have a negative baseline urine pregnancy test and agree to use a medically approved method of birth control for the duration of the study. All hormonal birth control must have been in use for a minimum of three months. Acceptable methods of birth control include:
   * Hormonal contraceptives including oral contraceptives, hormone birth control patch (Ortho Evra), vaginal contraceptive ring (NuvaRing), injectable contraceptives (Depo-Provera, Lunelle), or hormone implant (Norplant System)
   * Double-barrier method
   * Intrauterine devices
   * Non-heterosexual lifestyle or agrees to use contraception if planning on changing to heterosexual partner(s)
   * Vasectomy of partner at least 6 months prior to screening
3. Individuals with moderate stress as determined by a score of 14 - 26 on the Perceived Stress Scale
4. Agrees to maintain current sleep schedule throughout study
5. Must have a high school diploma or equivalent and basic computer skills
6. Agrees to avoid high caffeine consumption (examples include but not limited to no more than 2 cups/day of caffeinated coffee or tea)
7. Agrees to refrain from vigorous physical activity 24-hr prior to study visits
8. Agrees to maintain current lifestyle as much as possible including current sleep schedule until the end of the study
9. Willingness to complete questionnaires, records and diaries associated with the study, and to complete all clinic visits
10. Provided voluntary, written, informed consent to participate in the study
11. Healthy as determined by medical history, laboratory results, and as assessed by the QI

Exclusion Criteria:

1. Women who are pregnant, breastfeeding, or planning to become pregnant during the course of the trial
2. Participants who have a known allergy to the Investigational Product (IP) or Placebo active or inactive ingredients
3. Current employment that calls for rotating shift work or shift work that will disrupt normal circadian rhythm in the last 3 weeks
4. Travelled across 1 or more time zones in the 3 weeks prior to run-in and/or is anticipating more travel
5. Self-reported diagnosis with a stress or sleep disorder as assessed by the QI
6. Self-reported diagnosis of a neuropsychiatric and/or cognitive impairment as assessed by the QI
7. Self reported colour-blindness
8. Type I or Type II Diabetes
9. Unstable metabolic disease or chronic diseases as assessed by the QI
10. Current or history of any significant disease of the gastrointestinal tract as assessed by the QI
11. Unstable hypertension. Treatment on a stable dose of medication for at least 3 months will be considered by the QI
12. Significant cardiovascular event in the past 6 months as assessed by the QI
13. Major surgery in the past 3 months or individuals who have planned surgery during the course of the trial. Participants with minor surgery will be considered on a case-by-case basis by the QI
14. Cancer, except skin basal cell carcinoma completely excised with no chemotherapy or radiation with a follow up that is negative. Volunteers with cancer in full remission for more than five years after diagnosis are acceptable
15. Individuals with an autoimmune disease or are immune-compromised
16. History of or current diagnosis with kidney and/or liver diseases as assessed by the QI on a case-by-case basis, with the exception of history of kidney stones symptom-free for 6 months
17. Self reported current or pre-existing thyroid condition. Treatment on a stable dose of medication for at least 3 months will be considered by the QI
18. Self reported blood/bleeding disorders that will have an effect on safety outcomes as assessed by the QI
19. Self-reported alcohol or drug abuse within the last 12 months
20. High alcohol intake (>2 standard drinks per day)
21. Use of medicinal cannabinoid products, as assessed by the QI
22. Chronic use of cannabinoid products (≥2 times/week) and is unwilling to stop use for the duration of the study. Occasional use to be assessed by QI on a case-by-case basis
23. Use of tobacco and nicotine-containing products within 60 days of baseline and during the study period
24. Current use of prescribed medications which may affect stress, sleep, cognition, and/or mood (see Section 7.3.1)
25. Current use of over-the-counter medications, supplements, foods, and/or drinks which may affect stress, sleep, cognition, and/or mood unless willing to undergo the appropriate washout (see Section 7.3.2)
26. Clinically significant abnormal laboratory results at screening as assessed by the QI
27. Blood donation 30 days prior to baseline, during the study, or a planned donation within 30 days of the last study visit
28. Participation in other clinical research studies 30 days prior to baseline, as assessed by the QI
29. Individuals who are unable to give informed consent
30. Any other condition or lifestyle factor, that, in the opinion of the QI, may adversely affect the participant's ability to complete the study or its measures or pose significant risk to the participant

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2023-04-04 (Actual); Primary Completion 2023-07-17 (Actual); Study Completion 2023-07-17 (Actual)

PRIMARY OUTCOMES:
The difference in change in stress as assessed by salivary cortisol from baseline at Days 14 and 28 between AlphaWave® L-Theanine and Placebo. | Day 0, day 14, day 28

SECONDARY OUTCOMES:
The difference in change in stress as measured by the Perceived Stress Scale (PSS) from baseline at Days 14 and 28 between AlphaWave® L-Theanine and Placebo. | Day 0, day 14, day 28
The difference in change in the stress subscale as measured by the Depression Anxiety and Stress Scale (DASS)-21 from baseline at Days 14 and 28 between AlphaWave® L-Theanine and Placebo. | Day 0, day 14, day 28
The difference in change in the depression subscale as measured by the Depression Anxiety and Stress Scale (DASS)-21 from baseline at Days 14 and 28 between AlphaWave® L-Theanine and Placebo. | Day 0, day 14, day 28
The difference in change in the anxiety subscale as measured by the Depression Anxiety and Stress Scale (DASS)-21 from baseline at Days 14 and 28 between AlphaWave® L-Theanine and Placebo. | Day 0, day 14, day 28
The difference in change in the total score measured by the Depression Anxiety and Stress Scale (DASS)-21 from baseline at Days 14 and 28 between AlphaWave® L-Theanine and Placebo. | Day 0, day 14, day 28
The difference in change in sleep between AlphaWave® L-Theanine and Placebo from baseline at Days 14 and 28, as assessed by the Healthy People Sleep Quality Index (HPSQI). | Days 0, 14, and 28
The difference in change in sleep between AlphaWave® L-Theanine and Placebo from baseline at Days 14 and 28, as assessed by actigraphy readings. | Days 0, 14, and 28
  Actigraphy readings will include data on sleep duration, sleep onset, wake time, sleep latency, sleep efficiency, sleep stages, arousal count, and sleep score (0-100).
The difference in change in cognition between AlphaWave® L-Theanine and Placebo from baseline at Days 14 and 28. | Days 0, 14, and 28
  The difference in change in cognition will be assessed by the Computerized Mental Performance Assessment System (COMPASS): Stroop Test, Simple Reaction Time, and Choice Reaction Time.
The difference in change in mood between AlphaWave® L-Theanine and Placebo from baseline at Days 14 and 28. | Days 0, 14, and 28
  The difference in change in mood will be assessed by the Profile of Mood States (POMS) questionnaire.
Incidence of pre-emergent and post-emergent adverse events (AE) following supplementation with AlphaWave® L-Theanine and Placebo. | 28 days
Measurement of blood pressure (BP) following supplementation with AlphaWave® L-Theanine and Placebo. | screening, day 0, day 14, day 28
Measurement of heart rate (HR) following supplementation with AlphaWave® L-Theanine and Placebo. | screening, day 0, day 14, day 28
Measurement of aspartate aminotransferase (AST) following supplementation with AlphaWave® L-Theanine and Placebo. | screening, day 28
Measurement of alanine aminotransferase (ALT) following supplementation with AlphaWave® L-Theanine and Placebo. | screening, day 28
Measurement of alkaline phosphatase (ALP) following supplementation with AlphaWave® L-Theanine and Placebo. | screening, day 28
Measurement of total bilirubin following supplementation with AlphaWave® L-Theanine and Placebo. | screening, day 28
Measurement of creatinine following supplementation with AlphaWave® L-Theanine and Placebo. | screening, day 28
Measurement of electrolytes following supplementation with AlphaWave® L-Theanine and Placebo. | screening, day 28
  Electrolytes to be measured include sodium, potassium, and chloride.
Measurement of glucose following supplementation with AlphaWave® L-Theanine and Placebo. | screening, day 28
Measurement of estimated glomerular filtration rate (eGFR) following supplementation with AlphaWave® L-Theanine and Placebo. | screening, day 28
Measurement of white blood cell count (WBC) with differential following supplementation with AlphaWave® L-Theanine and Placebo. | screening, day 28
  WBC differentials include neutrophils, lymphocytes, monocytes, eosinophils, and basophils.
Measurement of red blood cell count (RBC) following supplementation with AlphaWave® L-Theanine and Placebo. | screening, day 28
Measurement of hemoglobin following supplementation with AlphaWave® L-Theanine and Placebo. | screening, day 28
Measurement of hematocrit following supplementation with AlphaWave® L-Theanine and Placebo. | screening, day 28
Measurement of platelet count following supplementation with AlphaWave® L-Theanine and Placebo. | screening, day 28
Measurement of immature granulocytes following supplementation with AlphaWave® L-Theanine and Placebo. | screening, day 28
Measurement of nucleated red blood cells (RBC) following supplementation with AlphaWave® L-Theanine and Placebo. | screening, day 28
Measurement of mean corpuscular volume (MCV) following supplementation with AlphaWave® L-Theanine and Placebo. | screening, day 28
Measurement of mean corpuscular hemoglobin (MCH) following supplementation with AlphaWave® L-Theanine and Placebo. | screening, day 28
Measurement of mean corpuscular hemoglobin concentration (MCHC) following supplementation with AlphaWave® L-Theanine and Placebo. | screening, day 28
Measurement of red blood cell distribution width (RDW) following supplementation with AlphaWave® L-Theanine and Placebo. | screening, day 28

CONTACTS AND LOCATIONS:
Overall Officials: David Crowley, MD, Principal Investigator — KGK Science Inc.
Locations (1):
- KGK Science Inc., London, Ontario, Canada

REFERENCES:
- [Derived] Moulin M, Crowley DC, Xiong L, Guthrie N, Lewis ED. Safety and Efficacy of AlphaWave(R) L-Theanine Supplementation for 28 Days in Healthy Adults with Moderate Stress: A Randomized, Double-Blind, Placebo-Controlled Trial. Neurol Ther. 2024 Aug;13(4):1135-1153. doi: 10.1007/s40120-024-00624-7. Epub 2024 May 17. PMID 38758503